CLINICAL TRIAL: NCT03315481
Title: Ultrasound Guided Repositioning of a New Suture-method Catheter for Adductor Canal Block - a Randomized Study in Healthy Volunteers
Brief Title: Ultrasound Guided Repositioning of a New Suture-Method Catheter for Adductor Canal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: H-16029530
Record Dates: First submitted 2017-03-01; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia; Pain, Postoperative; Pain; Pain, Joint
MeSH Terms: conditions — Pain, Postoperative; Pain; Arthralgia

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial in healthy volunteers. 12 volunteers will have suture-method catheters placed in the adductor canal of each leg using the long-axis plane and short-axis plane technique
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The volunteers are randomized using sealed opaque envelopes with a 1:1 ratio. The randomization defines which leg to be used for insertion of a catheter in the long-axis plane and which leg to be used for insertion in the short-axis plane of the adductor canal. Furthermore the randomization defines whether dislocation is executed in the direction of the entry or exit site. The envelopes are prepared by health personnel with no relation to the study and are based on a computer-generated randomization list.
  Investigator 2, evaluating loss of sensation to cold, will be blinded to insertion technique and direction of dislocation as well as assessments of spread within the adductor canal. Investigators 3+4 are blinded with regard to direction of dislocation, each other's assessment of spread and to assessments from investigator 1+2. They will be unblinded with regard to insertion technique when they perform US scans
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAX catheter insertion (Active Comparator): Ultrasound guided cather insertion in the short axis (SAX) of the adductor canal. Injection of lidocaine through the catheter
  Interventions: Procedure: SAX catheter insertion
- LAX catheter insertion (Active Comparator): Ultrasound guided cather insertion in the long axis (LAX) of the adductor canal. Injection of lidocaine through the catheter
  Interventions: Procedure: LAX catheter insertion

INTERVENTIONS:
Procedure: SAX catheter insertion — Suture-method catheter inserted in the short axis of the adductor canal
  Arms: SAX catheter insertion
Procedure: LAX catheter insertion — Suture-method catheter inserted in the long axis of the adductor canal
  Arms: LAX catheter insertion

SUMMARY:
This is a randomized clinical trial in healthy volunteers. 12 volunteers will have suture-method catheters placed in the adductor canal of each leg using the long-axis plane and short-axis plane technique. The investigators will inject LA in both catheters to confirm correct position. Following return of cold sensation the catheter is then displaced intentionally. The orifice is identified by injection of isotonic saline to ensure a proper displacement (spread outside of the adductor canal) and the distance from the delivery orifice of the catheter to the adductor canal is noted. A second investigator will assess distance from the LA delivery orifice of the catheter to the adductor canal using hydrodissection with isotonic saline to pinpoint the delivery orifice and subsequently reposition the catheter to obtain LA spread within the adductor canal. Successful repositioning is defined as a combination of LA spread within the adductor canal and loss of cold sensation on the medial part of the lower leg.

DETAILED DESCRIPTION:
The study objective is to investigate whether it is possible to reposition a displaced suture-method catheter using ultrasound.

A peripheral nerve catheter will be inserted on each side under US guidance. An investigator will insert one catheter in the short-axis plane of the adductor canal using an in plane technique: The needle is inserted through the vastus medialis into the adductor canal and exits superficial to the femoral artery through the sartorius muscle.

The second catheter is inserted from proximal to distal direction in the long-axis plane using a combination of in-plane and out-of-plane techniques.

10mL of isotonic saline is used for hydro-dissection for both catheter insertions to facilitate placement. Both catheters are injected with 15 mL LA with an immediate assessment of the spread being within or outside the adductor canal.

Loss of cold sensation in the cutaneous saphenous nerve innervation area will be evaluated 15 minutes after injection by another investigator, who is blinded to allocation and randomization.

Following return of normal sensory function the catheter is then intentionally displaced at least 2 cm outside the adductor canal in the direction of the entry or exit site according to randomization. The distance from the LA delivery orifice of the catheter to the adductor canal is noted. Adequate displacement requires that injection of isotonic saline does not result in spread within the adductor canal.

A third investigator will assess distance from the LA delivery orifice of the catheter to the adductor canal and subsequently reposition the catheter using saline to pinpoint location of the delivery orifice. Once the catheter is repositioned LA is injected. The US scan during LA injection is performed with a fourth investigator present to evaluate for satisfactory spread within the adductor canal. The 2 investigators will not communicate regarding the assessment of spread within the adductor canal.

Evaluation of cold sensation on the medial part of the lower leg is performed 15 minutes after 15mL LA (lidocaine 10 mg/mL) injection by investigator 2. The catheters are then removed and the study is completed.

Distance from catheter delivery orifices to the adductor canal is defined as following:

Distance from the LA delivery orifice to the fascia surrounding the adductor canal is noted in the short axis group. The distance from the LA delivery orifice to the penetration of the aponeurosis lying just below the sartorius muscle is noted in the long axis group. Both represent anatomical reference points for the adductor canal.

Satisfactory spread within the adductor canal is defined as following:

The LA injection spreads deeper along the lateral side of the femoral artery, observed in the two-dimensional plane while producing minimal displacement of the roof and the overlying sartorius muscle.

The injection may spread occasionally superficially over the femoral artery within the canal and will then force the artery deeper. If the injection spreads more medially and superficially over the saphenous nerve and femoral artery in an anterolateral to posteromedial direction, initially resembling the injections within the adductor canal but separates the sartorius muscle from the femoral artery by lifting the sartorius muscle medially off the hyperechoic roof of the adductor canal it is considered not to spread within the adductor canal.13

Successful primary placement and subsequent repositioning is defined as the combination of satisfactory spread within the adductor canal (assessed using SAX visualization of the adductor canal for both catheters) and loss of cold sensation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* ASA classification ≤ II.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Previous surgery or ongoing pain or other disability of investigated region resulting in sensory or neurologic deficits in the investigated region.
* Allergy to LA.
* Pregnancy (all female participants will be tested for urine hCG), breastfeeding, or unwilling to practice birth control during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Successful repositioning | 15 min after second injection
  Defined as a combination of spread within the adductor canal and loss of cold sensation on the medial part of the lower leg after repositioning and second LA injection.
  - investigator 3 will evaluate spread and investigator 2 will evaluate cold sensation

SECONDARY OUTCOMES:
Successful primary placement | 15 min after first injection
  Defined as a combination of spread within the adductor canal and loss of cold sensation after initial LA injection - investigator 1 will evaluate spread and investigator 2 will evaluate cold sensation
Estimation of Limits of Agreement | within 15 minutes, after displacement/repositioning.(recorded by after displacement and repeated just before attempted repositioning)
  in evaluation of displacement distance of the catheter between investigator 1 and 3
Interrater agreement for satisfactory spread within the adductor Canal, (Cohen's Kappa) | recorded immediately after second LA injection
  Investigator 3 and 4 will independently evaluate spread within the adductor canal.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias S Lyngeraa, MD, Principal Investigator — Research Unit, Department of Anaesthesiology and Intensive Care, Nordsjaellands Hospital Hilleroed
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jordahn ZM, Lyngeraa TS, Grevstad U, Rothe C, Lundstrom LH, Lange KHW. Ultrasound guided repositioning of a new suture-method catheter for adductor canal block - a randomized pilot study in healthy volunteers. BMC Anesthesiol. 2018 Oct 24;18(1):150. doi: 10.1186/s12871-018-0615-4. PMID 30355334